CLINICAL TRIAL: NCT07368335
Title: Efficacy and Safety of Endoscopic Treatment in Common Bile Duct Stone Based on the Electronic Endoscopic Surgery System: A Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Efficacy and Safety of a Novel ERCP Robot in the Treatment of Common Bile Duct Stone
Acronym: ERCP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0910-02; 20251106 (Other Grant/Funding Number: Shanghai Aohua Endoscopy Co., Ltd.)
Record Dates: First submitted 2026-01-06; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: ERCP; Robot Surgery; Common Bile Duct Stone
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional ERCP group (Active Comparator): This group will undergo conventional endoscopic common bile duct lithotomy with a regular electronic duodenoscope.
  Interventions: Device: Conventional ERCP
- Robotic-assisted ERCP group (Experimental)
  Interventions: Device: Robotic-assisted ERCP

INTERVENTIONS:
Device: Robotic-assisted ERCP — This group will receive endoscopic common bile duct lithotomy using the Electronic Endoscopic Surgery System produced by Shanghai Aohua Endoscopy Co., Ltd.
  Arms: Robotic-assisted ERCP group
Device: Conventional ERCP — This group will undergo conventional endoscopic common bile duct lithotomy with a regular electronic duodenoscope.
  Arms: Conventional ERCP group

SUMMARY:
Conventional endoscopic retrograde cholangiopancreatography (ERCP) is performed under fluoroscopic guidance, exposing endoscopists to ionizing radiation and posing risks of work-related musculoskeletal injury. Robotic-assisted ERCP may mitigate these occupational hazards and potentially enhance procedural precision and stability. However, robust clinical evidence regarding its performance and safety remains limited. This prospective, multicenter, randomized controlled non-inferiority trial is designed to evaluate the efficacy and safety of an ERCP robotic system (Electronic Endoscopic Surgery System) developed by Shanghai Aohua Photoelectricity Endoscope Co., Ltd. for common bile duct stone removal. A total of at least 200 subjects will be recruited and randomized 1:1 to either the experimental group or the control group. The experimental group will undergo robotic-assisted ERCP lithotomy using the aforementioned system, while the control group will receive conventional ERCP lithotomy using a standard duodenoscope.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years, inclusive.
2. Diagnosed with common bile duct stones based on symptoms, signs, laboratory tests, and imaging examinations, and deemed suitable by the investigator for endoscopic common bile duct stone removal (lithotomy).
3. Willing to comply with all study procedures; able to understand the study purpose, and voluntarily provide written informed consent.

Exclusion Criteria:

1. Severe cardiac, pulmonary, renal, or hepatic insufficiency, or mental disorders.
2. Active viral hepatitis.
3. Upper gastrointestinal stenosis, obstruction, or any condition preventing endoscopic access to the descending duodenum.
4. Known intolerance to anesthetics or hypersensitivity to contrast agents.
5. Non-lithogenic obstructive acute pancreatitis or acute exacerbation of chronic pancreatitis.
6. Pregnant or lactating women.
7. Active peptic ulcer or upper gastrointestinal hemorrhage within one month prior to informed consent.
8. Known severe bleeding tendency (coagulopathy).
9. History of upper gastrointestinal reconstruction surgery resulting in altered anatomy.
10. Previous endoscopic sphincterotomy of the duodenal papilla.
11. Inability to cooperate with ERCP procedures.
12. Participation in a drug clinical trial within the past 3 months, or in another medical device clinical trial (excluding non-interventional studies) within the past month.
13. Any other condition that, in the opinion of the investigator, may render the participant unsuitable for the trial (including but not limited to duodenal mucosal edema, papillary malformation, papillary surface ulcer, papillary fistula, or difficult-to-treat stones).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of bile duct stone extraction success | Baseline
  Stone extraction success was defined as complete clearance of the common bile duct during the same procedure.
Rate of adverse events | Through study completion, an average of 1 month

SECONDARY OUTCOMES:
Rate of biliary cannulation success | Baseline
  Biliary cannulation success was defined as achievement of deep biliary access.
Procedure time, including papilla localization time, cannulation time and stone extraction time | Baseline
  Papilla localization time was defined as the time required from insertion of the duodenoscope to accurate identification of the major duodenal papilla. Cannulation time was defined as the interval from first contact between the papilla and a wire-guided sphincterotome to successful deep biliary access. Stone extraction time was defined as the duration from successful biliary cannulation to complete stone removal, confirmed endoscopically and fluoroscopically. Total procedure time was measured from insertion of the duodenoscope into the esophagus to completion of all planned ERCP interventions.
Intraoperative radiation exposure time and radiation exposure dose of the principal operating investigator | Baseline
Success rate of external drainage | Baseline
Success rate of pancreatic duct stent placement | Baseline
Rate of intraoperative conversion | Baseline
  It is defined as the proportion of subjects who switched from endoscopic common bile duct lithotomy using the investigational device to other treatment modalities during the operation.
Evaluation of System Performance | Baseline
  The performance of the intraoperative investigational device was evaluated by the principal operating investigators using a three-grade rating system (Excellent, Good, Fair), following the procedures below:
  A three-grade rating system (Excellent, Good, Fair) was adopted for the evaluation. Three principal operating investigators from 3 clinical centers conducted independent evaluations based on the Evaluation Indicators and Criteria, respectively. The evaluation results are filled in the Evaluation Form for Surgical Procedure and Device Coordination.
Operational Comfort and Satisfaction Scores | Baseline
  This score is obtained through a questionnaire-based approach, and the questionnaire is designed to collect the comfort level and satisfaction degree ratings of the principal operating investigators (10 items in total).
  Each item is scored on a 1-5 scale, with scores ranging from 1 to 5 from left to right. The scoring definitions are as follows: 1 point for Strongly Agree; 2 points for Agree; 3 points for Neutral; 4 points for Disagree; 5 points for Strongly Disagree.
  A lower score indicates a better experience and higher satisfaction of the investigators with the use of the investigational device.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided